CLINICAL TRIAL: NCT00395018
Title: Study of the Antiviral Activity of Entecavir in Patients Receiving Liver Transplant Due to Chronic Hepatitis B Virus Infection
Brief Title: Antiviral Activity of Entecavir in Patients Receiving Liver Transplant Due to Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AI463-109
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B Virus, Liver Transplant
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- entecavir (Experimental)
  Interventions: Drug: entecavir

INTERVENTIONS:
Drug: entecavir — Tablets, Oral, 1 mg, once daily, up to 72 weeks
  Other Names: Baraclude; BMS-200475

SUMMARY:
The purpose of this clinical research study is to learn if the study drug entecavir will prevent the recurrence of hepatitis B virus (HBV) in participants who receive an orthotopic liver transplant (OLT) due to HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving orthotopic liver transplant (OLT) due to end-stage liver disease because of chronic HBV infection, with HBV-DNA < 172 IU/mL (approximately < 1000 copies/mL) prior to liver transplant
* Must have detectable hepatitis B surface antigen (HBsAg) at screening and for at least 24 weeks prior to screening

Exclusion Criteria:

* Patients with hepatocellular carcinoma with evidence of extrahepatic spread, multiple tumors ≥ 6.5 cm in diameter or there is up to three nodules ≥ 4.5 cm in diameter and total tumor diameter is ≥ 8 cm
* Co-infection with human immunodeficiency virus (HIV), cytomegalovirus (CMV), Epstein-Barr virus (EBV) or hepatitis C virus (HCV)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (9):
  - Northwestern University, Chicago, Illinois
  - Tulane University Hospital & Clinic, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - University Of Rochester Medical Center, Rochester, New York
  - University Of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
- Local Institution, Buenos Aires, Buenos Aires, Argentina
- Australia (2):
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Heidelberg, Victoria
- Brazil (3):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- France (3):
  - Local Institution, Clichy
  - Local Institution, Paris
  - Local Institution, Villejuif
- Italy (3):
  - Local Institution, Bologna
  - Local Institution, Roma
  - Local Institution, Torrette Di Ancona
- Local Institution, Seoul, South Korea
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia
- Taiwan (2):
  - Local Institution, Kaohsiung City
  - Local Institution, Taipei

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 109 participants were enrolled at 27 investigative sites.
Pre-assignment Details: Of the 109 participants enrolled, 65 were treated and 61 received therapy for at least 1 month. Of the 44 participants who were never treated, 23 no longer met study criteria, 9 due to administrative reason by sponsor, 6 withdrew consent, 3 due to other reasons, 2 died, 1 due to poor/non-compliance.
Groups:
- Entecavir (ETV): ETV tablets, Oral, 1.0 mg, once daily, up to 72 weeks
Period: On-Treatment
Arm/Group | Entecavir (ETV)
Started | 65 (Started = treated (participants who received at least 1 dose of study therapy))
DISCONTINUED PRIOR TO WEEK 72 VISIT | 10
DISCONTINUED AT OR AFTER WEEK 72 VISIT | 0
Completed | 55 ("Completed" means received treatment through Week 72)
Not Completed | 10
Not completed — Death | 4
Not completed — Other Reason | 2
Not completed — Poor/non-compliance | 2
Not completed — Subject no longer meets study criteria | 2
Period: Off-Treatment Follow-up
Arm/Group | Entecavir (ETV)
Started | 5 (Treated participants who discontinued =<72 weeks and did not start other anti-HBV therapy)
Completed | 1 ("Completed" means completed the study)
Not Completed | 4
Not completed — Followup no longer required per protocol | 1
Not completed — Lost to Follow-up | 2
Not completed — Poor/non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 65
Age Continuous [Median (Full Range); unit: years] | 51.0 [23 to 68]
Age, Customized [Number; unit: participants]
  21-64 years | 60
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 24
  Black/African American | 7
  Native Hawaiian/Other Pacific Islander | 1
  White | 25
  Other | 8
Race/Ethnicity, Customized [Number; unit: participants] — Participants in United States of America (USA) only.
  participants
    Hispanic/Latino | 0
    Not Hispanic/Latino | 14
Region of Enrollment [Number; unit: participants]
  Argentina | 2
  Australia | 5
  Brazil | 12
  France | 12
  Italy | 6
  Korea, Republic of | 7
  Spain | 3
  Taiwan | 4
  United States | 14
HBV DNA by PCR [Median (Full Range); unit: log10 IU/mL] | 0.8 [0.8 to 3.7]
Hepatitis B Surface Antigen [Number; unit: participants]
  Positive | 61
  Negative | 4
Hepatitis B E Antigen (HBeAg) [Number; unit: participants]
  Positive | 7
  Negative | 58
Hepatitis B E Antibody (HBeAb) [Number; unit: participants]
  Positive | 48
  Negative | 17
International Normalized Ratio [Median (Full Range); unit: ratio] — Evaluated in 63 participants at baseline.
  ratio | 1.51 [0.86 to 7.10]
Albumin [Median (Full Range); unit: g/dL] | 3.0 [1.8 to 4.7]
Alanine Aminotransferase (ALT) [Median (Full Range); unit: U/L] | 43 [10 to 1485]
Total Bilirubin [Median (Full Range); unit: mg/dL] | 2.4 [0.2 to 31.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBV Deoxyribonucleic Acid (DNA) => 50 IU/mL by Polymerase Chain Reaction (PCR) at Week 72
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan High+Pure system (HPS) assay. HBV DNA => 50 IU/mL = approximately => 300 copies/mL.
Time Frame: At 72 weeks
Population: Evaluable population: Treated participants who received at least 1 month of ETV therapy. Last observation carried forward (LOCF) approach was used for participants with no measurement in the specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 61
percentage of participants | 0 [0.0 to 5.9]

2. Secondary Outcome: Distribution of ALT Levels Through 72 Weeks: Overall
Description: ALT is an enzyme present in serum and various tissues of the body, associated commonly with the liver. Elevated levels of ALT often suggests existence of medical problems which includes viral hepatitis. Normal range varies from laboratory to laboratory. Values of 5-60 U/L is usually considered normal. ALT abnormality = >1.25 x ULN (upper limit of normal).
Time Frame: On Day 1 (baseline) and at week 4, 12, 24, 36, 48, 60, 72
Population: Evaluable population: Treated participants who received at least 1 month of ETV therapy.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 61
U/L
  Baseline | 158.7 (36.20)
  Week 4 | 61.2 (10.12)
  Week 12 | 28.4 (2.66)
  Week 24 (n=59) | 28.4 (3.37)
  Week 36 (n=58) | 41.2 (8.20)
  Week 48 (n=57) | 24.9 (1.91)
  Week 60 (n=53) | 30.6 (4.04)
  Week 72 (n=54) | 26.9 (2.81)

3. Secondary Outcome: Percentage of Participants With HBV DNA < 50 IU/mL (Approximately 300 Copies/mL) by PCR at the End of Post-dosing Follow-up
Description: HBV DNA assessments were to be performed using the Roche COBAS® TaqMan AmpliPrep assay. HBV DNA < 50 IU/mL = approximately 300 copies/mL.
Time Frame: At 72 weeks + 24 weeks follow-up
Population: This analysis was planned if > 10% of treated participants had HBV DNA measurements during the off-treatment follow-up period.
Measure: Number; unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With HBeAg Loss at Week 72 (for HBeAg-positive Participants)
Description: HBeAg is a hepatitis B viral protein. HBeAg loss = HBeAg-negative at the specified analysis week.
Time Frame: At week 72
Population: HBeAg positive participants at baseline who received at least 1 month of ETV therapy. LOCF approach was used for participants with no measurement in the specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 7
percentage of participants | 100 [59.0 to 100.0]

5. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 72 (for HBeAg-positive Participants)
Description: HBeAg is a hepatitis B viral protein. HBeAg Seroconversion = HBeAg Loss and Presence of Hepatitis B e Antibody (HBeAb).
Time Frame: At week 72
Population: HBeAg-positive participants at baseline who received at least 1 month of ETV therapy. LOCF approach was used for participants with no measurement in the specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 7
percentage of participants | 0 [0.0 to 41.0]

6. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 72
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is an early marker of infection. HBsAg loss = HBsAg-negative at the specified analysis week.
Time Frame: At week 72
Population: Evaluable participants: Treated participants who received at least 1 month of ETV therapy. LOCF approach was used for participants with no measurement in the specified visit window.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 61
percentage of participants | 96.7 [88.7 to 99.6]

7. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 72
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is an early marker of infection. HBs seroconversion is defined as HBsAg loss with positive HBsAb.
Time Frame: At week 72
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 61
percentage of participants | 80.3 [68.2 to 89.4]

8. Secondary Outcome: Percentage of Participants With HBsAg Recurrence At Week 72
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is an early marker of infection. HBsAg recurrence is defined as having detectable HBsAg among participants who have already experienced loss of HBsAg on-treatment. HBsAg recurrence = HBsAg-positive at the specified analysis week.
Time Frame: At week 72
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 61
percentage of participants | 3.3 [0.4 to 11.3]

9. Secondary Outcome: Total Bilirubin at Week 72
Description: Bilirubin measures are used to diagnose or monitor liver functioning or diseases that include hepatitis. Viral hepatitis is one of the condition in which bilirubin levels are elevated. Normal range varies from laboratory to laboratory. Bilirubin abnormality : => 1.1 x ULN mg/dL.
Time Frame: At week 72
Population: Treated participants with measures available at week 72.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 54
mg/dL | 0.79 (0.079)

10. Secondary Outcome: Prothrombin Time (PT) at Week 72
Description: Prothrombin, a liver protein, plays an important role in the extrinsic pathway of clotting. Increased prothrombin time indicates abnormal liver functioning. Normal prothrombin time varies from laboratory to laboratory. Generally, normal prothrombin time varies between 10 to 13.2 seconds. Abnormal PT: > 1.01 x ULN.
Time Frame: At week 72
Population: Treated participants with measures available at week 72.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 53
seconds | 13.32 (0.305)

11. Secondary Outcome: Number of Participants With Liver Rejection Through Week 72
Time Frame: Through week 72
Population: Treated participants: Participants who received atleast 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 65
participants | 18

12. Secondary Outcome: Number of Participants With Re-transplantation Through Week 72
Time Frame: Through week 72
Population: Treated population: Participants who received atleast 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 65
participants | 3

13. Secondary Outcome: Participants With Adverse Events (AE), Serious Adverse Events (SAE), and Discontinuations From Study Drug Due to AEs (On-treatment [OT] and Off-treatment Follow-up [OF])
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or an overdose. Toxicity grading by modified WHO grade system. Grade (GR) 2=moderate; GR3=severe; GR4=very severe. OT=from start of dosing to end of dosing+5 days; OF=from end of dosing+6 days to start of other anti-HBV therapy or end of follow-up.
Time Frame: OT:From start of dosing through Week 72 + 5 days; OF:End of OT through 24-weeks follow-up
Population: Treated population: Participants who received atleast 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 65
participants
  Death-OT | 4
  SAEs-OT | 36
  SAEs-OF (n=5) | 0
  Discontinuation due to AEs-OT | 0
  Any AE-OT | 62
  Any AE-OF (n=5) | 0
  Related AEs-OT | 11
  Grade 2 - 4 related AEs-OT | 8
  Grade 3 - 4 AEs-OT | 30

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities On-treatment (OT) and Off-Treatment Follow-up(OF): Hematology (All Grades)
Description: Criteria for hematology abnormalities were: Hemoglobin : <11.0 g/dL; White Blood Cells : <4000/mm^3; Neutrophils : <1500/mm^3; Platelets : < 99,000/mm^3; International Normalized Ratio (INR) : increase >= 0.5 from baseline.
Time Frame: OT:From start of dosing through Week 72 + 5 days; OF:End of OT through 24-weeks follow-up
Population: Treated population: All subjects who received atleast 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 65
participants
  HEMOGLOBIN-OT | 56
  HEMOGLOBIN-OF (n=5) | 1
  WHITE BLOOD CELLS-OT | 50
  WHITE BLOOD CELLS-OF (n=5) | 2
  NEUTROPHILS (Includes absolute bands)-OT | 24
  NEUTROPHILS (Includes absolute bands)-OF (n=5) | 1
  PLATELETS-OT | 40
  PLATELETS-OF (n=5) | 2
  INR-OT (n=63) | 30
  INR-OF (n=4) | 0

15. Secondary Outcome: Number of Participants With Laboratory Abnormalities On-treatment (OT) and Off-Treatment (OF) Follow-up: Serum Chemistry (All Grades)
Description: Normal ranges are local lab data and vary according to the site. Criteria for laboratory abnormalities:ALT:>1.25xULN;AST:>1.25xULN;ALP:>1.25xULN;Total Bilirubin:>1.1xULN;Serum Lipase:>1.10xULN;Creatinine:>1.1xULN;Blood Urea Nitrogen:>1.25xULN;Hyperglycemia:>116mg/dL;Hypoglycemia:<64mg/dL;Hyponatremia:<132meq/L;Hypernatremia:>148meq/L;Hypokalemia:<3.4meq/L;hyperkalemia:>5.6meq/L;Hypochloremia:<93meq/L;Hyperchloremia:>113meq/L;Albumin: Decrease >= 1g/dL from baseline and < 3 g/dL. HYPER=value>ULN(upper limit of normal). HYPO=value<LLN (lower limit of normal).
Time Frame: OT:From start of dosing through Week 72 + 5 days; OF:End of OT through 24-weeks follow-up
Population: Treated population: Participants who received atleast 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 65
participants
  ALANINE AMINOTRANSFERASE (ALT)-OT | 54
  ALT-OF (n=4) | 0
  ASPARTATE AMINOTRANSFERASE (AST)-OT | 56
  AST-OF (n=4) | 0
  ALKALINE PHOSPHATASE (ALP)-OT | 34
  ALP-OF (n=4) | 1
  ALBUMIN-OT (n=64) | 51
  ALBUMIN-OF (n=3) | 0
  TOTAL BILIRUBIN-OT | 57
  TOTAL BILIRUBIN-OF (n=4) | 0
  SERUM LIPASE-OT (n=64) | 37
  SERUM LIPASE-OF (n=3) | 1
  CREATININE-OT | 43
  CREATININE-OF (n=4) | 0
  BLOOD UREA NITROGEN-OT | 43
  BLOOD UREA NITROGEN-OF (n=4) | 0
  HYPERGLYCEMIA-OT (n=64) | 52
  HYPERGLYCEMIA-OF (n=3) | 0
  HYPOGLYCEMIA-OT (n=64) | 15
  HYPOGLYCEMIA-OF (n=3) | 0
  HYPERNATREMIA-OT | 7
  HYPERNATREMIA-OF (n=4) | 0
  HYPONATREMIA-OT | 14
  HYPONATREMIA-OF (n=4) | 0
  HYPERKALEMIA-OT | 15
  HYPERKALEMIA-OF (n=4) | 0
  HYPOKALEMIA-OT | 22
  HYPOKALEMIA-OF (n=4) | 0
  HYPERCHLOREMIA-OT | 11
  HYPERCHLOREMIA-OF (n=4) | 0
  HYPOCHLOREMIA-OT | 7
  HYPOCHLOREMIA-OF (n=4) | 0

16. Primary Outcome: Number of Participants With HBV DNA by PCR >= 50 IU/mL Through Week 72
Description: as for outcome 1
Time Frame: At baseline (day 1), week 12, 24, 36, 48, 60, and 72
Population: Evaluable population: Treated participants who received at least 1 month of ETV therapy. Non-Completer = Missing (NC = M) approach was used where participants who discontinued early or were missing the measurement were excluded from the specific analysis.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Entecavir (ETV)
Number analyzed (Participants) | 61
participants
  Baseline | 3 [1.0 to 13.7]
  Week 12 (n = 54) | 0 [0.0 to 6.6]
  Week 24 (n = 58) | 0 [0.0 to 6.2]
  Week 36 (n = 10) | 0 [0.0 to 30.8]
  Week 48 (n = 49) | 0 [0.0 to 7.3]
  Week 60 (n = 48) | 0 [0.0 to 7.4]
  Week 72 (n = 49) | 0 [0.0 to 7.3]

ADVERSE EVENTS:
Time Frame: From start of dosing through Week 72 + 5 days
Arm/Group | Entecavir (ETV)
Serious Adverse Events (participants affected / at risk) | 36/65
Other Adverse Events (participants affected / at risk) | 58/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir (ETV) (N=65)
Aspartate aminotransferase increased (Investigations) | 2
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1
Biliary dilatation (Hepatobiliary disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Haematoma infection (Infections and infestations) | 1
Renal failure acute (Renal and urinary disorders) | 3
Septic shock (Infections and infestations) | 1
Shock haemorrhagic (Vascular disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 2
Biliary fistula (Hepatobiliary disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Intra-abdominal haemorrhage (Vascular disorders) | 1
Liver transplant rejection (Immune system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Device related infection (Infections and infestations) | 1
Hepatic artery thrombosis (Hepatobiliary disorders) | 3
Meningitis aseptic (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Wound infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Eye infection toxoplasmal (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Vision blurred (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Arterial rupture (Vascular disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Hepatic artery stenosis (Hepatobiliary disorders) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatitis B virus test (Investigations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyrexia (General disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vein disorder (Vascular disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Biliary tract disorder (Hepatobiliary disorders) | 1
Hernial eventration (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Transplant rejection (Immune system disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Multi-organ failure (General disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir (ETV) (N=65)
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 15
Hypoaesthesia (Nervous system disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Bile duct stenosis (Hepatobiliary disorders) | 5
Constipation (Gastrointestinal disorders) | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 8
Headache (Nervous system disorders) | 13
Liver function test abnormal (Investigations) | 6
Overweight (Metabolism and nutrition disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 4
Depression (Psychiatric disorders) | 4
Renal impairment (Renal and urinary disorders) | 4
Tremor (Nervous system disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 4
Vomiting (Gastrointestinal disorders) | 9
Anaemia (Blood and lymphatic system disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Catheter site discharge (General disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 4
Incision site pain (Injury, poisoning and procedural complications) | 4
Nausea (Gastrointestinal disorders) | 8
Procedural pain (Injury, poisoning and procedural complications) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 10
Hypertension (Vascular disorders) | 22
Insomnia (Psychiatric disorders) | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 17
Hypokalaemia (Metabolism and nutrition disorders) | 4
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 4
Sepsis (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.